CLINICAL TRIAL: NCT03894800
Title: Determination of Analgesic Equipotent Doses of Inhaled Metoxyflurane vs. Intravenous Fentanyl Using Cold Pressor Test (CPT) in Volunteers: A Randomized, Double Blind, Placebo-controlled Crossover Study.
Brief Title: Determination of Analgesic Equipotent Doses of Inhaled Metoxyflurane vs. Intravenous Fentanyl
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Harald Lenz, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-0910-3; 2018-003939-30 (EudraCT Number)
Record Dates: First submitted 2019-03-04; First posted 2019-03-29 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Acute Pain; Trauma; Hypovolemia
Keywords: metoxyflurane; pain; fentanyl; cold pressor test
MeSH Terms: conditions — Acute Pain; Wounds and Injuries; Hypovolemia; Pain | interventions — Methoxyflurane; Fentanyl

STUDY DESIGN:
Intervention Model Description: This is a randomized, double blind, placebo-controlled crossover study.
Who Masked: Participant, Investigator
Masking Description: Labeling of the IMPs will be done by one a nurse anesthetist not participating in the study. The study drugs, will be distributed in a pre-packed in identical, opaque envelopes (the same day as the drugs will be used). The envelopes are not to be broken until randomization of the patient is done
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Methoxyflurane (M) (Active Comparator): A session starts with a CPT - cold pressor test (time -15 minutes). Then a 10 minutes rest before the subject receives a syringe of NaCl intravenous (time -5 minutes). At the same time the subject begin to inhale metoxyflurane through the inhalator. The subject should first take 10 breath through the inhalator. This will take approximately 1-1.5 minutes. The subject then take a break, and then inhale the rest of the dosage before time zero.
  At time zero a new CPT will be performed. At time 15 minutes the last CPT will be performed.
  The subjects will undergo CPT (cold pressor test) to determine the analgesic effect of the drugs. Each test lasts up to 90 seconds and endpoints are NRS scores every 10 second.
  Interventions: Drug: Methoxyflurane (M); Drug: NaCl (C)
- Fentanyl (F1) (Active Comparator): A session starts with a CPT (time -15 minutes). Then a 10 minutes rest before the subject receives a syringe of fentanyl 0.025 mg intravenous (time -5 minutes). At the same time the subject begin to inhale NaCl through the inhalator. The subject should first take 10 breath through the inhalator. This will take approximately 1-1.5 minutes. The subject then take a break, and then inhale the rest of the dosage before time zero.
  At time zero a new CPT will be performed. At time 15 minutes the last CPT will be performed.
  The subjects will undergo CPT (cold pressor test) to determine the analgesic effect of the drugs.Each test lasts up to 90 seconds and endpoints are NRS scores every 10 second.
  Interventions: Drug: Fentanyl (F1); Drug: NaCl (C)
- Fentanyl (F2) (Active Comparator): A session starts with a CPT (time -15 minutes). Then a 10 minutes rest before the subject receives a syringe of fentanyl 0.05 mg intravenous (time -5 minutes). At the same time the subject begin to inhale NaCl through the inhalator. The subject should first take 10 breath through the inhalator. This will take approximately 1-1.5 minutes. The subject then take a break, and then inhale the rest of the dosage before time zero.
  At time zero a new CPT will be performed. At time 15 minutes the last CPT will be performed.
  The subjects will undergo CPT (cold pressor test) to determine the analgesic effect of the drugs. Each test lasts up to 90 seconds and endpoints are NRS scores every 10 second.
  Interventions: Drug: Fentanyl (F2); Drug: NaCl (C)
- NaCl (C) (Placebo Comparator): A session starts with a CPT (time -15 minutes). Then a 10 minutes rest before the subject receives a syringe of NaCl intravenous (time -5 minutes). At the same time the subject begin to inhale NaCl through the inhalator. The subject should first take 10 breath through the inhalator. This will take approximately 1-1.5 minutes. The subject then take a break, and then inhale the rest of the dosage before time zero.
  At time zero a new CPT will be performed. At time 15 minutes the last CPT will be performed.
  The subjects will undergo CPT (cold pressor test) to determine the analgesic effect of the drugs. Each test lasts up to 90 seconds and endpoints are NRS scores every 10 second.
  Interventions: Drug: NaCl (C)

INTERVENTIONS:
Drug: Methoxyflurane (M) — The subjects will undergo CPT (cold pressor test) to determine the analgesic effect of the drugs, in this intervention inhalation of metoxyflurane 3 ml and NaCl i.v. will be administered.(13,14) The CPT will be conducted using a temperature-controlled bath with circulating 3°C water (FP 45-HE Refrigerated/Heating Circulator, Julabo Labortechnic, 77960 Seelback, Germany). The subjects submerge their right hand to the wrist with fingers abducted for up to 90 s. The endpoints are NRS scores every 10 s.This test will be performed 3 times for each session.
  Other Names: NaCl
  Arms: Methoxyflurane (M)
Drug: Fentanyl (F1) — The subjects will undergo CPT (cold pressor test) to determine the analgesic effect of the drugs, in this intervention fentanyl 0.025 mg i.v. and NaCl for inhalation will be administered(13,14) The CPT will be conducted using a temperature-controlled bath with circulating 3°C water (FP 45-HE Refrigerated/Heating Circulator, Julabo Labortechnic, 77960 Seelback, Germany). The subjects submerge their right hand to the wrist with fingers abducted for up to 90 s. The endpoints are NRS scores every 10 s.This test will be performed 3 times for each session.
  Other Names: NaCl (C)
  Arms: Fentanyl (F1)
Drug: Fentanyl (F2) — The subjects will undergo CPT (cold pressor test) to determine the analgesic effect of the drugs, in this intervention fentanyl 0.05 mg i.v. and NaCl for inhalation will be administered.(13,14) The CPT will be conducted using a temperature-controlled bath with circulating 3°C water (FP 45-HE Refrigerated/Heating Circulator, Julabo Labortechnic, 77960 Seelback, Germany). The subjects submerge their right hand to the wrist with fingers abducted for up to 90 s. The endpoints are NRS scores every 10 s.This test will be performed 3 times for each session.
  Other Names: NaCl (C)
  Arms: Fentanyl (F2)
Drug: NaCl (C) — The subjects will undergo CPT (cold pressor test) to determine the analgesic effect of the drugs, in this intervention NaCl i.v. and NaCl inhal will be used - placebo(13,14) The CPT will be conducted using a temperature-controlled bath with circulating 3°C water (FP 45-HE Refrigerated/Heating Circulator, Julabo Labortechnic, 77960 Seelback, Germany). The subjects submerge their right hand to the wrist with fingers abducted for up to 90 s. The endpoints are NRS scores every 10 s.This test will be performed 3 times for each session.

SUMMARY:
The aim of this study is to determinate the equipotent doses of inhaled metoxyflurane vs. intravenous fentanyl.

DETAILED DESCRIPTION:
Traumatized patients frequently experience pain prehospital due to the fear of adverse cardiovascular effects (e.g. hypotension) and respiration depression of opioid treatment, leading to insufficient analgesia. Therefore, there is of interest to investigate other analgesics that do not have these adverse effects.

In Norway, methoxyflurane has been approved for the emergency relief of moderate to severe trauma pain in conscious adult patients. Metoxyflurane (Penthrox®) do not have these adverse effects (hypotension and respiration depression). It is easy to administrate via an inhalator, and is therefore suitable for use prehospital. This would possible help to treat pain better prehospital.

There exists no data of how effective metoxyflurane is as an analgesic compared to an opioid. The aim of this study is to determinate the equipotent doses of inhaled metoxyflurane vs. intravenous fentanyl.

Ten healthy volunteers (18 - 64 years) will be enrolled in a randomized, double blind, placebo-controlled, crossover study using a standard experimental pain model: CPT- Cold pressor test (ice water). Our group has used this experimental pain model in earlier studies and a crossover study is suitable to compare different drugs.

Possible side effects will be recorded for both metoxyflurane and fentanyl: sedation, dizziness, itching, nausea and vomiting. Respiration frequency and non-invasive blood pressure will be recorded every as possible low blood pressure or respiration depression can occur.

The aim of this study is to determinate equipotent doses of inhaled metoxyflurane vs. intravenous fentanyl. We have chosen to compare with fentanyl (the comparator) because it is a well-known drug in clinical practice for acute pain treatment. In addition, both drugs have a fast onset (minutes) and the analgesic effect last for approximately the same time interval (20-30 min). Therefore, they are comparable in a clinical setting.

There exists no exact data of equipotent doses between metoxyflurane and fentanyl, only retrospective clinical data. One retrospective study compared intranasal fentanyl with inhaled metoxyflurane for visceral pain prehospital in 1024 patients. The initial dose of fentanyl was 0.018 mg and the total mean dose at hospital arrival was 0.036 mg. In the metoxyflurane group 51.9% received 3 ml, a second dose was used in 41.9% and 6.2% received a third dose. Metoxyflurane produced the greatest initial pain scores reduction, and intranasal fentanyl provided greater pain reduction by hospital arrival.

From these data we have chosen two doses of fentanyl to be compared with 3 ml Penthrox: 0.025 mg and 0.05 mg intravenous. Both drugs will also be compared to placebo (NaCl 9 mg/ml).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers
2. Age 18 - 64
3. Both sex
4. No chronic disease
5. No regular medication
6. Recruited from the general population
7. Signed informed consent and expected cooperation of the subjects for the treatment and follow up must be obtained and documented according to ICH GCP, and national/local regulations

Exclusion Criteria:

1. Use of pain medication the last 2 days before a session
2. Use of complementary medicine the last 2 days before a session
3. Use of regular medication
4. Previous substance abuse
5. Pregnancy
6. Know allergies or serious side effects to opioids or metoxyflurane
7. Use of alcohol last 24 h before each session
8. Exclusion criteria with respect to fentanyl:
9. Hypersensitivity opposite the active substance (fentanyl) or other opioids
10. Hypersensitivity opposite the excipients (to fentanyl): sodiumclorid, water for injection, hydrochloric acid or sodium hydroxide
11. Respiratory depression without artificial ventilation
12. Use of MAO-inhibitor or use of MAO-inhibitor by two weeks before inclusion
13. Elevated intracranial pressure or brain trauma
14. Hypovolemia or hypotension
15. Myasthenia gravis
16. Exclusion criteria with respect to metoxyflurane:
17. Use metoxyflurane as anesthetic
18. Hypersensitivity opposite metoxyflurane or fluorinated anesthetics
19. Hypersensitivity opposite the excipient (to metoxyflurane):

    Butylhydroksytoulen
20. Malignant hyperthermia or persons with suspect genetic predisposition for malignant hyperthermia
21. History (to the volunteer or family) of serious adverse effects after administration of inhalation anesthetics
22. Volunteers showing sign of liver damage after use of metoxyflurane or halogenated anesthetics
23. History of liver disease
24. Clinical significant reduced kidney function or history of kidney disease
25. Changed of level of consciousness of any cause, including brain trauma, drugs or alcohol
26. Clinical detected cardiovascular unstability
27. Clinical detected respiratory depression

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2019-10-29 (Actual)

PRIMARY OUTCOMES:
NRS (numeric rating scale) scores during the second CPT, which starts 5 minutes after drug administration and lasts for 90 seconds. NRS is a scale from 0 to 10 (0, 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10). 0 = no pain and 10 = worst pain imaginable. | 90 seconds
  NRS (numeric rating scale) scores during CPT (Cold pressor test) 5 minutes after drug administration. The CPT lasts for 90 seconds. The endpoints are NRS scores every 10. second during the CPT.

SECONDARY OUTCOMES:
NRS (numeric rating scale) scores during the second CPT, which starts 20 minutes after drug administration and lasts for 90 seconds. This is a scale from 0 to 10 (0, 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10). 0 = no pain and 10 = worst pain imaginable. | 90 seconds
  NRS scores during CPT (Cold pressor test) 20 minutes after drug administration (15 minutes after last CPT).The CPT lasts for 90 seconds. The endpoints are NRS scores every 10. second during the CPT.

CONTACTS AND LOCATIONS:
Overall Officials: Harald Lenz, Phd, Principal Investigator — Oslo University Hospital
Locations (1):
- Harald Lenz, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Albrecht E, Taffe P, Yersin B, Schoettker P, Decosterd I, Hugli O. Undertreatment of acute pain (oligoanalgesia) and medical practice variation in prehospital analgesia of adult trauma patients: a 10 yr retrospective study. Br J Anaesth. 2013 Jan;110(1):96-106. doi: 10.1093/bja/aes355. Epub 2012 Oct 11. PMID 23059961
- [Result] Neighbor ML, Honner S, Kohn MA. Factors affecting emergency department opioid administration to severely injured patients. Acad Emerg Med. 2004 Dec;11(12):1290-6. doi: 10.1197/j.aem.2004.07.014. PMID 15576519
- [Result] Stephen CR. Clinical applications of methoxyflurane. Acta Anaesthesiol Scand Suppl. 1966;24:215-22. doi: 10.1111/j.1399-6576.1966.tb01127.x. No abstract available. PMID 6003600
- [Result] Mazze RI. Methoxyflurane revisited: tale of an anesthetic from cradle to grave. Anesthesiology. 2006 Oct;105(4):843-6. doi: 10.1097/00000542-200610000-00031. PMID 17006084
- [Result] Grindlay J, Babl FE. Review article: Efficacy and safety of methoxyflurane analgesia in the emergency department and prehospital setting. Emerg Med Australas. 2009 Feb;21(1):4-11. doi: 10.1111/j.1742-6723.2009.01153.x. PMID 19254307
- [Result] Rosen M, Latto P, Asscher AW. Kidney function after methoxyflurane analgesia during labour. Br Med J. 1972 Jan 8;1(5792):81-3. doi: 10.1136/bmj.1.5792.81. PMID 5007074
- [Result] Clark RB, Beard AG, Thompson DS. Renal function in newborns and mothers exposed to methoxyflurane analgesia for labor and delivery. Anesthesiology. 1979 Nov;51(5):464-6. doi: 10.1097/00000542-197911000-00020. No abstract available. PMID 496064
- [Derived] Lenz H, Hoiseth LO, Comelon M, Draegni T, Rosseland LA. Determination of equi-analgesic doses of inhaled methoxyflurane versus intravenous fentanyl using the cold pressor test in volunteers: a randomised, double-blinded, placebo-controlled crossover study. Br J Anaesth. 2021 May;126(5):1038-1045. doi: 10.1016/j.bja.2020.12.045. Epub 2021 Mar 4. PMID 33676727

DOCUMENTS (2):
  • Informed Consent Form (2019-03-07): https://cdn.clinicaltrials.gov/large-docs/00/NCT03894800/ICF_001.pdf
  • Study Protocol and Statistical Analysis Plan (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/00/NCT03894800/Prot_SAP_002.pdf